CLINICAL TRIAL: NCT00810511
Title: Evaluation of Two Silicone Hydrogel Lenses Over a One Month Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-335-C-007
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2012-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lotrafilcon A (Experimental): Investigational, spherical, silicone hydrogel contact lenses
  Interventions: Device: Lotrafilcon A contact lens
- Comfilcon A (Active Comparator): Commercially marketed, spherical, silicone hydrogel contact lenses
  Interventions: Device: Comfilcon A contact lens

INTERVENTIONS:
Device: Lotrafilcon A contact lens — Silicone hydrogel contact lens
  Arms: Lotrafilcon A
Device: Comfilcon A contact lens — Silicone hydrogel contact lens
  Arms: Comfilcon A

SUMMARY:
The purpose of this trial is to compare two different contact lenses during 4 weeks of wear.

ELIGIBILITY:
Inclusion Criteria:

* Current soft contact lens wearer who wear their habitual lenses for no less than 10 hours a day, 5 days a week
* Have a need for correction in both eyes and be correctable to at least 20/40 distance vision in each eye while wearing trial lenses
* Replace lenses on a weekly or longer schedule
* Other protocol inclusion/exclusion criteria may apply

Exclusion Criteria:

* Requires concurrent ocular medication
* Eye injury or surgery within twelve weeks immediately prior to enrollment
* Evidence of systemic or ocular abnormality, infection, or disease likely to affect successful wear of contact lenses or use of their accessory solutions
* Current soft toric lens wearers
* Those who dispose of their soft lenses on a daily basis
* Current NIGHT & DAY® or Biofinity® lens wearers
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lotrafilcon A | Comfilcon A
Started | 107 | 106
Completed | 97 | 102
Not Completed | 10 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 9 | 1
Not completed — death in the family | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — deposits on contact lens | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lotrafilcon A | Comfilcon A | Total
Number analyzed (Participants) | 107 | 106 | 213
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 10 | 21
  Between 18 and 65 years | 96 | 96 | 192
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (9.8) | 31.8 (11.0) | 31.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 84 | 168
  Male | 23 | 22 | 45
Region of Enrollment [Number; unit: participants]
  United States | 107 | 106 | 213

OUTCOME MEASURES:

1. Primary Outcome: Comfort at End of Day
Description: Evaluated by the subject as a single, retrospective evaluation of 4-week wear time. Measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: After 4 weeks of wear
Population: One subject in the Lotrafilcon A arm was excluded from efficacy analysis due to a protocol deviation.
Measure: Mean (Standard Deviation); unit: Scale of 1-10
Arm/Group | Lotrafilcon A | Comfilcon A
Number analyzed (Participants) | 96 | 102
Scale of 1-10 | 6.5 (2.4) | 6.9 (2.4)

ADVERSE EVENTS:
Time Frame: 8 weeks, duration of the study
Arm/Group | Lotrafilcon A | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/106
Other Adverse Events (participants affected / at risk) | 0/107 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.